CLINICAL TRIAL: NCT04977713
Title: Effects of Acupressure and Shower Applied in the Delivery on the Intensity of Labor Pain and Postpartum Comfort
Brief Title: Delivery Pain and Postpartum Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KırklareliAS-4
Record Dates: First submitted 2021-06-25; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Labor Pain; Hydrotherapy; Acupressure; Postpartum Period
Keywords: labor pain; shower; acupressure; midwife; postpartum comfort
MeSH Terms: conditions — Labor Pain | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: The randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure group (Experimental): In the acupressure uterine contractions were checked before the care application began. Acupressure was applied when the women's cervical dilation reached 4-5 cm, 6-7 cm and 8-10 cm. This method was applied 18 times during uterine contractions. The application stopped at the end of each contraction and resumed once another contraction started. No application was performed between contractions.
  Interventions: Other: Acupressure
- Shower Group (Experimental): The shower group, uterine contractions were checked before the care application began. A shower was applied when the women's cervical dilation reached 4-5 cm, 6-7 cm and 8-10 cm. This method was applied 18 times during uterine contractions. The application stopped at the end of each contraction and resumed once another contraction started. No application was performed between contractions.
  Interventions: Other: Shower
- Control group (No Intervention): The women in the control group underwent routine hospital care. They were administered neither pharmacological nor nonpharmacological methods to reduce labour pain.

INTERVENTIONS:
Other: Acupressure — A researcher sat behind the women to comfortably access the sacral area and be in the appropriate position. The researcher then applied deep rotational pressure on the BL32 points until her nail bed colour changed to prevent any discomfort in the participants
  Arms: Acupressure group
Other: Shower — During uterine contractions, these participants took a shower while standing, with a researcher on hand to assist her (average time: 20 minutes). The water's temperature was between 22°C and 26°C.
  Arms: Shower Group

SUMMARY:
In this study was aimed that acupressure applied on the BL32 point and shower application reduced the intensity of labor pain experienced by the pregnant women in the active phase of labor and increased their postpartum comfort

DETAILED DESCRIPTION:
Acupressure and shower are methods that can help reduce pain severity. This study thus aims to determine the effects of acupressure and shower on labour pain and postpartum comfort. This study was a randomized controlled trial (RCT). This study was the control group consisted of 40 pregnant women, while the experimental groups (acupressure and shower) consisted of 80 pregnant women in total. The experimental groups received routine labour care and either acupressure or showers upon reaching three cervical dilations (4-5, 6-7 and 8-10 cm). The control group only received routine labour care. A maternal information form (MIF), the Visual Analog Scale for Pain (VASP) and the Postpartum Comfort Questionnaire (PPCQ) were used to collect data. CONSORT checklist was used to report the current study.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were being 20-40 years of age;
* Having a foetus in vertex presentation
* Having a foetus weighing 2.5-4 kg, as determined through ultrasonography
* Being primiparous
* Being between 37 and 42 gestational weeks with a single foetus
* Having planned to have a spontaneous vaginal delivery
* Not having used nonpharmacological pain control methods previously
* Having a cervical dilation less than 5 cm (Dabiri et al., 2014)
* Not having received analgesia or anaesthesia.

Exclusion Criteria:

* Were having a systemic disease during pregnancy (gestational diabetes, hypertension)
* Taking medication regularly
* Having a problem that prevented the woman from communicating
* Undergoing psychiatric treatment (pharmacotherapy or psychotherapy)
* Requiring an operative vaginal delivery (forceps, vacuum)
* Receiving pharmacological interventions for labour pain.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 120 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Reduce labor pain | Evaluation was done until delivery (on average between 8-12 hours)
  The participants were applicated acupressure, and shower as for birth pain. Pain has been evaluated with VASP.
Postpartum comfort levels | 2 hours after birth
  Postpartum comfort levels of the groups who received acupressure and shower in the postpartum period were evaluated.Postpartum comfort level has been evaluated with PPCQ.
A maternal information form | before birth
  This form consisted of 13 items asking for the participants' sociodemographic characteristics
Visual Analog Scale for Pain (VASP) | Evaluation was done until delivery (on average between 8-12 hours)
  This scale is a 0-10 cm ruler developed by Bond and Pilowsky (Hawker et al., 2011; Aslan and Öztürk, 2014; Kömürcü and Ergin, 2014; Bond and Pilowsky, 1996). VASP is a 10 cm ruler which assessment with "no pain" at one end and "worst pain" at the other end. A Turkish validity and reliability study of the VASP was performed by Aslan and Öztürk (Aslan and Öztürk, 2014; Kömürcü and Ergin, 2014; Aslan, 2004).
Postpartum Comfort Questionnaire (PPCQ) | 2 hours after birth
  The 48-item General Comfort Scale, developed by Kolcaba (Kolcaba, 1994), was first adapted into Turkish in 2008 by Kuğuoğlu and Karabacak, who also conducted a Turkish validity and reliability study on the scale (Kuğuoğlu and Karabacak, 2008). Based on the Turkish version of the GCS, Karakaplan and Yıldız (Karakaplan and Yıldız, 2010) developed the PPCQ. The PPCQ is a 5-point questionnaire with 34 items. Participants give items between 1 (strongly agree) and 5 points (strongly disagree). The lowest score possible is 34, and the highest score is 170, with higher scores indicating higher comfort levels.
Evalution labour pain | Evaluation was done until delivery (on average between 8-12 hours)
  VASP was evaluated before and after acupressure and shower applications.
Evalution postpartum comfort | 2 hours after birth
  Postpartum Comfort levels were evaluated in the postpartum period.

CONTACTS AND LOCATIONS:
Overall Officials: AYCA SOLT KIRCA, Phd, Principal Investigator — Kırklareli University; DERYA KANZA GÜL, Md, Phd, Principal Investigator — Medipol University
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No